CLINICAL TRIAL: NCT01232049
Title: A Randomized, Open-label, Multiple Dose, Crossover Study to Evaluate a Pharmacokinetic Drug Interaction and Safety Between Pitavastatin and Valsartan in Healthy Male Subjects
Brief Title: Drug Interaction and Safety Between Pitavastatin and Valsartan (CWP-PTV-101)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: JW Pharmaceutical (Industry)
Responsible Party: ChoongWae Parma Corporation, Clinical Research Team
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2010-0577
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2010-10

CONDITIONS: Healthy
Keywords: healthy volunteers
MeSH Terms: interventions — pitavastatin; Valsartan

ARMS (3):
- A (Experimental): Pitavastatin 4mg
  Interventions: Drug: Multiple Oral Dose of
- B (Experimental): Valsartan 320mg
  Interventions: Drug: Multiple Oral Dose of
- C (Experimental): Pitavastatin 4mg + Valsartan 320mg
  Interventions: Drug: Multiple Oral Dose of

INTERVENTIONS:
Drug: Multiple Oral Dose of — Pitavastatin 4mg
  Other Names: Livalo®
  Arms: A; C
Drug: Multiple Oral Dose of — Valsartan 320mg
  Other Names: Diovan®
  Arms: B; C

SUMMARY:
This study is designed to evaluate a pharmacokinetic drug interaction and safety between Pitavastatin and Valsartan in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Adult males aged 20 to 50 years at screening.
* No significant congenital/chronic disease. No symptoms in physical examination.
* Appropriate subjects as determined by past medical history, laboratory tests, serology and urinalysis.
* Be able to understand the objective, method of the study, the characteristics of investigational drug, and comply with the requirement of the study. Subject must provide written informed consent prior to study participation.

Exclusion Criteria:

* History or presence of liver, kidney, or nervous system disease, respiratory disorders, endocrinological disorders, hemato-oncologic, cardiovascular or psychiatric or cognitive disorders.
* History of gastrointestinal disorders (bleeding, ulceration, hemorrhoids, piles) or disorders of absorption, distribution, metabolism, excretion.
* History of known hypersensitivity to drugs including valsartan and pitavastatin.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Safety (normal results for safety tests) | 39days
  Adverse events Physical examination, vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Kyun-Seop Bae, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Jung JA, Noh YH, Jin S, Kim MJ, Kim YH, Jung JA, Lim HS, Bae KS. Pharmacokinetic interaction between pitavastatin and valsartan: a randomized, open-labeled crossover study in healthy male Korean volunteers. Clin Ther. 2012 Apr;34(4):958-65. doi: 10.1016/j.clinthera.2012.01.026. Epub 2012 Mar 10. PMID 22410289
- See also: Clinical Research Center, Asan Medical Center — http://crc.amc.seoul.kr